CLINICAL TRIAL: NCT07179913
Title: The Improvement of Low-dose Esketamine on Postoperative Depression in Patients Undergoing Bariatric Surgery With Preoperative Depression:A Prospective Radomized Controlled Trial
Brief Title: The Improvement of Low-dose Esketamine on Postoperative Depression in Patients Undergoing Bariatric Surgery With Preoperative Depression
Acronym: esketamine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, lizhiwen, study director, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 25K322-001
Record Dates: First submitted 2025-09-03; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Depressed; Bariatric Surgery
Keywords: esketamine; bariatric surgery; depression
MeSH Terms: conditions — Consciousness Disorders; Depression | interventions — Esketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine (Placebo Comparator)
  Interventions: Drug: Dexmedetomidine
- esketamine (Experimental)
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — For the subjects in the experimental group, esketamine 50mg/2ml was diluted with normal saline up to 50ml (with a concentration of esketamine at 1mg/ml), anesthesia induction begins with intravenous infusion of esketamine 0.25mg/kg (0.375ml/kg•h drug preparation solution), with a pumping duration of 40 minutes.After the operation, esketamine 0.25mg/kg and sufentanil 1.5ug/kg were added to the postoperative analgesic pump dilute to 100ml with normal saline, with a background dose of 2ml/h and a single booster dose of 2ml.
  Arms: esketamine
Drug: Dexmedetomidine — For the control group subjects, dexmedetomidine at a dose of 0.2mg/2ml was diluted with normal saline up to 50ml(dexmedetomidine concentration of 4μg/ml), anesthesia induction begins with intravenous infusion of 0.5μg/kg (0.083ml/kg•h), with a pumping duration of 40 minutes. The postoperative analgesic pump was added after the operation dilute with normal saline at a dose of 0.5μg/kg of dexmedetomidine and 1.5 μg/kg of sufentanil 100ml, with a background dose of 2ml/h and a single booster dose of 2ml.
  Arms: dexmedetomidine

SUMMARY:
The aim of this study is to observe the antidepressant effect of low-dose esketamine in obese patients with preoperative depression and seeking bariatric surgery. We speculate that intraoperative infusion and the addition of a small dose of esketamine to the postoperative analgesic pump can help reduce the proportion of patients with depression after surgery, and may further improve postoperative recovery, reduce the use of postoperative opioids, shorten postoperative hospital stay, and improve postoperative quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and <65 years old
* Patients with a BMI greater than 35 kg/m^2
* Hamilton Depression score ≥7 points
* Planned to undergo elective laparoscopic sleeve gastrectomy

Exclusion Criteria:

* ASA ≥ grade IV
* Those who have had or are currently suffering from mental disorders other than anxiety and depression, such as schizophrenia, bipolar disorder, organic mental disorders, etc.
* Those who are unable to cooperate in completing the scale assessment
* Have received ketamine/esketamine treatment, or are allergic to ketamine/esketamine
* Clarify ischemic cardiomyopathy or severe liver and kidney dysfunction (Child pugh grade C, CKD stage G5)
* People with opioid dependence and those who have been taking various types of painkillers for a long time (more than 3 months)
* Participate in other research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale ≥7 | Seven days after the operation
  The proportion of patients with depression (Hamilton Depression score ≥7)

SECONDARY OUTCOMES:
the proportion of patients with depression | 30 days, 3 months, 6 month and 1 year after the operation
  The proportion of patients with depression

OTHER OUTCOMES:
BMI in kg/m^2 | 30 days, 3 months, 6 months and 1 year after operation
  BMI in kg/m^2
the proportion of patients with anxeity | 30 days, 3 months, 6 months and 1 yea rafter operation
  the proportion of patients with anxeity
living quality score | 30 days, 3 months, 6 months and 1 year after operation
  living quality score

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwen Li, Doctor of Medicine, Study Director — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: Yes